CLINICAL TRIAL: NCT01572480
Title: Carfilzomib, Lenalidomide, and Dexamethasone in High-Risk Smoldering Multiple Myeloma: a Clinical and Correlative Pilot Study
Brief Title: Carfilzomib, Lenalidomide, and Dexamethasone for Smoldering Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elizabeth Hill, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120107; 12-C-0107
Record Dates: First submitted 2012-04-05; First posted 2012-04-06 (Estimated); Results first posted 2022-09-13 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Proteasome Inhibitor; Immunomodulatory Agents; Combination Therapy; Anti-Myeloma Activity
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A - (closed) - Carfilzomib with Revlimid and Dexamethasone (Experimental): Carfilzomib (intravenous (IV), Days 1, 2, 8, 9, 15, and 16 of the 28-day cycle); Revlimid (by mouth (PO), Days 1-21 of the 28-day cycle; exception: not given on cycle 1 day 1); and Dexamethasone (PO or IV, Days 1, 2, 8, 9, 15, 16, 22, and 23 of the 28-day cycle; exception: not given on cycle 1 day 1)
  Interventions: Drug: Carfilzomib; Drug: Revlimid; Drug: Dexamethasone
- Group B - Carfilzomib with Revlimid and Dexamethasone (Experimental): Carfilzomib (intravenous (IV), Days 1, 2, 8, 9, 15, and 16 of the 28-day cycle); Revlimid (by mouth (PO), Days 1-21 of the 28-day cycle); and Dexamethasone (PO or IV, Days 1, 2, 8, 9, 15, 16, 22, and 23 of the 28-day cycle)
  Interventions: Drug: Carfilzomib; Drug: Revlimid; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib intravenous (IV) 20-36 mg/m^2 per dose on days 1, 2, 8, 9, 15, and 16 of each cycle based on arm; until disease progression or unacceptable toxicity.
  Other Names: Kyprolis
Drug: Revlimid — Revlimid by mouth (PO) 25 mg/day, days 1-21 every 28 days of each cycle based on arm; until disease progression or unacceptable toxicity.
  Other Names: Lenalidomide
Drug: Dexamethasone — Dexamethasone by mouth (PO) 20 mg per dose on days 1, 2, 8, 9, 15, 16, 22, and 23 of each cycle based on arm; until disease progression or unacceptable toxicity.
  Other Names: Ozurdex

SUMMARY:
Background:

* Multiple myeloma is a blood cancer that affects the plasma cells. These cells help produce antibodies and fight infection. Smoldering multiple myeloma (SMM) is a related condition that may develop into multiple myeloma. The current standard of care for SMM is close follow-up without treatment until multiple myeloma develops. However, researchers are studying possible treatments for SMM itself. One possible treatment involves a combination of cancer treatment drugs.
* Lenalidomide is a drug that may help reduce or prevent the growth of cancer cells. Dexamethasone is a steroid that is often given with other anti-cancer drugs. These two drugs are an approved treatment for multiple myeloma that has not responded to at least one other treatment. Carfilzomib is an experimental drug that has been effective in treating multiple myeloma. Researchers want to combine these three drugs to see if they are a safe and effective treatment for SMM.

Objectives:

- To see if carfilzomib, lenalidomide, and dexamethasone are a safe and effective treatment for smoldering multiple myeloma.

Eligibility:

- Individuals at least 18 years of age who have SMM that is likely to progress to multiple myeloma.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests, and baseline bone marrow scans. Bone marrow samples will also be collected.
* Participants will have eight 28-day cycles of treatment with the three study drugs. The drugs will be given as tablets or as infusions. Treatment will be monitored with frequent blood tests and study visits.
* After the first four cycles, participants who are eligible for a stem cell transplant will have their stem cells collected and stored for future use.
* At the end of eight cycles, participants whose disease has not progressed will have up to 12 more cycles of treatment with lenalidomide tablets alone.

DETAILED DESCRIPTION:
Background:

Smoldering multiple myeloma (SMM) is a precursor condition to multiple myeloma (MM) defined by the clinical parameters of M-protein >= 3.0 g/dL or bone marrow plasma cells >= 10% and absence of end organ disease.

Risk of progression of high risk SMM at 5 years is 72-75% with median time to progression < 2 years.

The current standard of care for SMM is close follow-up without treatment until symptomatic MM develops. However, International Myeloma Working Group (IMWG) states "Preventive clinical trials need to be considered for patients with high risk smoldering myeloma".

Carfilzomib is a new proteasome inhibitor with potent anti-MM effects

Objectives:

To assess the response rate of cyclophosphamide, lenalidomide, and dexamethasone (CRd) in patients with high-risk SMM, focusing on the

Minimal residual disease (MRD(-) Complete Response (CR) rate

Eligibility:

SMM according to the International Myeloma Working Group definition; i.e.:

Serum M-protein >=3 g/dl and/or bone marrow plasma cells >=10 % and < 60%

Absence of anemia: Hemoglobin >10 g/dl

Absence of renal failure: serum creatinine < 2.0 mg/dL.

Absence of hypercalcemia: Calcium (Ca) < 10.5 mg/dl or 2.65 mmol/L

Absence of lytic bone lesion

Involved/un-involved light chain ratio must be < 100

Measurable disease

High-risk SMM per Mayo Clinic, Spanish Programa de Estudio y Tratamiento de las Hemopatías Malignas (PETHEMA), or the Rajkumar, Landgren, Mateos criteria

Age >=18 years

Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Adequate laboratory parameters as defined in the protocol

Design:

Single arm pilot trial of combination therapy (carfilzomib, lenalidomide, and dexamethasone) for high risk smoldering multiple myeloma

Patients will receive 8 cycles of induction combination therapy of CRd

Each cycle consists of 28-days

After 4 cycles of therapy, transplant eligible patients may choose to undergo stem cell collection

After 8 cycles of CRd, patients will receive lenalidomide extended dosing (phase I) for 12 cycles. After 12 cycles, patients will have the option to continue extended dosing (phase II) for one additional year.

Patients will have routine blood work with serum protein electrophoresis (SPEP) and free light chains monthly during the induction phase. Laboratory evaluations may be spread out to every 3 months during the maintenance and follow-up phases.

Pre-treatment, post-treatment and follow-up bone marrow biopsies will be obtained for confirmation of diagnosis, response and correlative studies

Patients will also undergo evaluation for minimal residual disease at regular interval time points, using multi-parametric flow cytometry and fluorodeoxyglucose (FDG)-positron emission tomography (PET)-computed tomography (CT)

This single arm pilot study will plan on initially enrolling 12 evaluable patients to detect a very good partial response (VGPR) from baseline. A replicate cohort of 16 evaluable patients will then be enrolled in order to more precisely define the response rate to the CRd regimen in this population. Accrual will then be extended to a total of 50 evaluable patients in order to estimate the MRD(-) CR rate with reasonable precision. To allow for a number of inevaluable patients and screen failures, the accrual ceiling will be set at 63.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histologically or cytologically confirmed Smoldering Multiple Myeloma confirmed by the Laboratory of Pathology, national Cancer Institute (NCI) or the Department of Laboratory Medicine, Clinical Center (CC) based on the International Myeloma Working Group Criteria:

* Serum M-protein greater than or equal to 3 g/dl and/or bone marrow plasma cells greater than or equal 10% and <60%
* Absence of anemia: Hemoglobin >10 g/dl
* Absence of renal failure: serum creatinine < 2.0 mg/dL
* Absence of hypercalcemia: Calcium (Ca) <10.5 mg/dl
* Absence of lytic bone lesion on X-ray, computed tomography (CT), or positron-emission tomography (PET)/CT and not more than 1 lesion on spinal magnetic resonance imaging (MRI). (NOTE: At the discretion of the investigator, PET/CT may replace MRI in patients who have a contraindication to MRI.)
* Involved-un-involved light chain ratio must be <100

Measurable disease within the past 4 weeks defined by any one of the following:

* Serum monoclonal protein greater than or equal to 1.0 g/dl
* Urine monoclonal protein >200 mg/24 hour
* Serum immunoglobulin free light chain >10 mg/dL AND abnormal kappa/lambda ratio

NOTE: As of Amendment L (version date 05/17/2018), the primary endpoint is minimal residual disease (MRD(-) Complete Response (CR) rate; therefore, per the discretion of the Principal Investigator, patients without measurable disease (e.g., M-spike <1) may also be enrolled. This is in line with the most recent International Myeloma Working Group (IMWG) multiple myeloma (MM) response criteria.

Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of carfilzomib in combination with lenalidomide in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.

Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).

Patients must have normal organ and marrow function as defined below:

- absolute neutrophil count (ANC) greater than or equal to1.0 K/uL

NOTE: At the discretion of the investigator, patients with an ANC of 0.5 K/uL <1.0 K/uL may also be enrolled if clinically appropriate (e.g., patients with a baseline neutropenia that is chronic and that does not cause complications)

* platelets greater than or equal to 75 K/uL
* hemoglobin greater than or equal to 8 g/dL(transfusions are permissible)
* total bilirubin less than or equal to 1.5 times institutional upper limit of normal
* aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) less than or equal to 3.0 times institutional upper limit of normal
* Serum creatinine less than or equal to 1.5 X institutional ULN. If serum creatinine is above 1.5 X ULN, Creatinine Clearance (CrCl) or estimated glomerular filtration rate (eGFR) (estimated glomerular filtration rate) must be greater than or equal to 50 ml/min.

  * Creatinine clearance (CrCl) will be calculated by Cockcroft-Gault method. CrCl (calculated) = (140 - Age) x Mass (in kilograms) x [0.85 if Female] 72 x Serum Creatinine (in mg/dL).
  * eGFR will be calculated by either of the following well established formulas: modification of diet in renal disease (MDRD) or the chronic kidney disease (CKD)-epidemiology collaboration (EPI) (institutional standard) equations
* CrCl may also be determined by measuring a 24 hour urine collection. The measured CrCl must be greater than or equal to 50 ml/min.

In addition to having Smoldering Multiple Myeloma (SMM), patients must also be classified as 'high-risk SMM' per Mayo Clinic or Spanish Programa de Estudio y Tratamiento de las Hemopatías Malignas (PETHEMA) criteria.

Criteria set forward by Rajkumar, Landgren, Mateos[14] may also be used to define high risk disease, namely clonal bone marrow plasma cells greater than or equal to 10% and any one or more of the following:

* Serum M protein greater than or equal to 30g/L
* Immunoglobulin A (IgA) SMM
* Immunoparesis with reduction of 2 uninvolved immunoglobulin isotypes
* Serum involved/uninvolved free light chain (FLC) ratio greater than or equal to 8 (but less than 100)
* Progressive increase in M protein level (evolving type of SMM; increase in serum M protein by greater than or equal to 25% on 2 successive evaluations within a 6-month period)
* Clonal bone marrow plasma cells (BMPCs) 50%-60%
* Abnormal plasma cells (PCs) immunophenotype (greater than or equal to 95% of BMPCs are clonal) and reduction of greater than or equal to 1 uninvolved immunoglobulin isotypes
* t(4;14) or del(17p) or 1q gain
* Increased circulating PCs
* MRI with diffuse abnormalities or 1 focal lesion
* PET-CT with focal lesion with increased uptake without underlying osteolytic bone destruction

All study participants must be registered into the mandatory RevAssist program and be willing and able to comply with the requirements of Risk Evaluation and Mitigation Strategy (REMS).

The effects of carfilzomib and lenalidomide on the developing human fetus are unknown. The immunomodulatory agents used in this trial (i.e., lenalidomide) are known to be teratogenic. Women of childbearing potential and men must agree to use adequate contraception. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.

Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. In regard to carfilzomib, FCBP and their male partners must agree to use at least one method of effective contraception for at least 30 days after the

last dose of carfilzomib and males must agree to use contraception and not to donate sperm for at least 90 days after the last dose of carfilzomib.

Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients who are receiving any other investigational agents.

Concurrent systemic treatment or prior therapy within 4 weeks for SMM

- Treatment with corticosteroids for other indications is permitted

Patients with a diagnosis of MM as defined by the 2014 IMWH diagnostic criteria.

Contraindication to any concomitant medication, including antivirals, anticoagulation prophylaxis, tumor lysis prophylaxis, or hydration given prior to therapy

History of allergic reactions attributed to compounds of similar chemical or biologic composition to carfilzomib or lenalidomide agents used in study, such as bortezomib or thalidomide, in addition to patients with known allergy to sulfobutyl ether <=- cyclodextrin (Captisol).

Uncontrolled hypertension or diabetes

Pregnant or lactating females. Pregnant women are excluded from this study. The effects of carfilzomib on a developing human fetus are unknown. Lenalidomide is teratogenic with unknown potential for abortifacient effects. Breastfeeding women and women planning on breastfeeding may not participate. No studies of carfilzomib have been conducted on breast feeding women and it is not known if it is excreted in milk. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Carfilzomib/Lenalidomide, breastfeeding should be discontinued if the mother is treated with Carfilzomib/Lenalidomide.

Significant cardiovascular disease with New York Heart Association (NYHA) Class II, III or IV symptoms, or hypertrophic cardiomegaly, or restrictive cardiomegaly, or myocardial infarction within 3 months prior to enrollment, or unstable angina, or unstable arrhythmia

Active hepatitis B or C infection

Has refractory gastrointestinal (GI) disease with refractory nausea/vomiting, inflammatory bowel disease, or bowel resection that would prevent absorption

Significant neuropathy >Grade 2 at the time of first dose or within 14 days of enrollment.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations within 2 weeks that would limit compliance with study requirements.

History of other malignancy (apart from basal cell carcinoma of the skin, or in situ cervix carcinoma) except if the patient has been free of symptoms and without active therapy during at least 2 years or if, at the clinical discretion of the investigator, the risks of this study do not outweigh the potential benefits on a case to case basis.

Major surgery within 1 month prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hill, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Background] Perez-Persona E, Vidriales MB, Mateo G, Garcia-Sanz R, Mateos MV, de Coca AG, Galende J, Martin-Nunez G, Alonso JM, de Las Heras N, Hernandez JM, Martin A, Lopez-Berges C, Orfao A, San Miguel JF. New criteria to identify risk of progression in monoclonal gammopathy of uncertain significance and smoldering multiple myeloma based on multiparameter flow cytometry analysis of bone marrow plasma cells. Blood. 2007 Oct 1;110(7):2586-92. doi: 10.1182/blood-2007-05-088443. Epub 2007 Jun 18. PMID 17576818
- [Background] Dispenzieri A, Kyle RA, Katzmann JA, Therneau TM, Larson D, Benson J, Clark RJ, Melton LJ 3rd, Gertz MA, Kumar SK, Fonseca R, Jelinek DF, Rajkumar SV. Immunoglobulin free light chain ratio is an independent risk factor for progression of smoldering (asymptomatic) multiple myeloma. Blood. 2008 Jan 15;111(2):785-9. doi: 10.1182/blood-2007-08-108357. Epub 2007 Oct 17. PMID 17942755
- [Background] Kyle RA, Durie BG, Rajkumar SV, Landgren O, Blade J, Merlini G, Kroger N, Einsele H, Vesole DH, Dimopoulos M, San Miguel J, Avet-Loiseau H, Hajek R, Chen WM, Anderson KC, Ludwig H, Sonneveld P, Pavlovsky S, Palumbo A, Richardson PG, Barlogie B, Greipp P, Vescio R, Turesson I, Westin J, Boccadoro M; International Myeloma Working Group. Monoclonal gammopathy of undetermined significance (MGUS) and smoldering (asymptomatic) multiple myeloma: IMWG consensus perspectives risk factors for progression and guidelines for monitoring and management. Leukemia. 2010 Jun;24(6):1121-7. doi: 10.1038/leu.2010.60. Epub 2010 Apr 22. PMID 20410922
- [Derived] Kazandjian D, Diamond B, Papadimitriou M, Hill E, Sklavenitis-Pistofidis R, Ziccheddu B, Blaney P, Chojnacka M, Durante M, Maclachlan K, Young R, Usmani S, Davies F, Getz G, Ghobrial I, Korde N, Morgan G, Maura F, Landgren O. Genomic Profiling to Contextualize the Results of Intervention for Smoldering Multiple Myeloma. Clin Cancer Res. 2024 Oct 1;30(19):4482-4490. doi: 10.1158/1078-0432.CCR-24-0210. PMID 38652812
- [Derived] Kazandjian D, Hill E, Dew A, Morrison C, Roswarski J, Korde N, Emanuel M, Petrosyan A, Bhutani M, Calvo KR, Dulau-Florea A, Kwok M, Lee MJ, Lee S, Lindenberg L, Mailankody S, Manasanch E, Maric I, Mena E, Patel N, Tageja N, Trepel JB, Turkbey B, Wang HW, Wang W, Yuan C, Zhang Y, Braylan R, Choyke P, Stetler-Stevenson M, Steinberg SM, Figg WD Sr, Roschewski M, Landgren O. Carfilzomib, Lenalidomide, and Dexamethasone Followed by Lenalidomide Maintenance for Prevention of Symptomatic Multiple Myeloma in Patients With High-risk Smoldering Myeloma: A Phase 2 Nonrandomized Controlled Trial. JAMA Oncol. 2021 Nov 1;7(11):1678-1685. doi: 10.1001/jamaoncol.2021.3971. PMID 34529025
- [Derived] Bhutani M, Turkbey B, Tan E, Korde N, Kwok M, Manasanch EE, Tageja N, Mailankody S, Roschewski M, Mulquin M, Carpenter A, Lamping E, Minter AR, Weiss BM, Mena E, Lindenberg L, Calvo KR, Maric I, Usmani SZ, Choyke PL, Kurdziel K, Landgren O. Bone marrow abnormalities and early bone lesions in multiple myeloma and its precursor disease: a prospective study using functional and morphologic imaging. Leuk Lymphoma. 2016 May;57(5):1114-21. doi: 10.3109/10428194.2015.1090572. Epub 2016 Apr 7. PMID 26690712
- [Derived] Korde N, Roschewski M, Zingone A, Kwok M, Manasanch EE, Bhutani M, Tageja N, Kazandjian D, Mailankody S, Wu P, Morrison C, Costello R, Zhang Y, Burton D, Mulquin M, Zuchlinski D, Lamping L, Carpenter A, Wall Y, Carter G, Cunningham SC, Gounden V, Sissung TM, Peer C, Maric I, Calvo KR, Braylan R, Yuan C, Stetler-Stevenson M, Arthur DC, Kong KA, Weng L, Faham M, Lindenberg L, Kurdziel K, Choyke P, Steinberg SM, Figg W, Landgren O. Treatment With Carfilzomib-Lenalidomide-Dexamethasone With Lenalidomide Extension in Patients With Smoldering or Newly Diagnosed Multiple Myeloma. JAMA Oncol. 2015 Sep;1(6):746-54. doi: 10.1001/jamaoncol.2015.2010. PMID 26181891
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0107.html

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Carfilzomib (intravenous (IV), Days 1, 2, 8, 9, 15, and 16 of the 28-day cycle); Revlimid (by mouth (PO), Days 1-21 of the 28-day cycle; exception: not given on cycle 1 day 1); and Dexamethasone (PO or IV, Days 1, 2, 8, 9, 15, 16, 22, and 23 of the 28-day cycle; exception: not given on cycle 1 day 1)
  Carfilzomib intravenous (IV) 20-36 mg/m^2 per dose on days 1, 2, 8, 9, 15, and 16 of each cycle based on arm; until disease progression or unacceptable toxicity.
  Revlimid by mouth (PO) 25 mg/day, days 1-21 every 28 days of each cycle based on arm; until disease progression or unacceptable toxicity.
Period: Participants Enrolled
Arm/Group | All Participants
Started | 55
Completed | 54
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Drug Administration
Arm/Group | All Participants
Started | 54
Completed | 53 (2 participants discontinued drug administration early because of adverse events, thus 1 was taken off study and 1 proceeded to maintenance.)
Not Completed | 1
Not completed — Discontinued drug/Off Study | 1
Period: Initiated Maintenance Therapy
Arm/Group | All Participants
Started | 53
Completed | 50
Not Completed | 3
Not completed — Discontinued maintenance therapy/experienced adverse events and withdrew consent | 1
Not completed — Discontinued maintenance therapy/experienced adverse events | 2
Period: Completed Maintenance Therapy
Arm/Group | All Participants
Started | 50
Completed | 30
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.83 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 38
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Northeast | 20
  United States: Southeast | 28
  United States: Southwest | 2
  United States: West | 4
  United States: Missing | 1
Cytogenetic Risk Group [Count of Participants; unit: Participants] — High risk cytogenetics was defined as del17p,t(14;16), t(14;20), and 1q gain. These cytogenetic abnormalities identified by fluorescence in situ hybridization (FISH) confer a worse prognosis. Per the International Myeloma Working Group (IMWG), participants with high risk cytogenetics may have impaired response to treatment and worse overall survival (OS).
  Participants
    High Risk | 20
    Standard Risk | 27
    Unknown | 7
Myeloma-defining event per International Myeloma Working Group (IMWG) 2014 [Number; unit: events] — This trial was for high risk smoldering myeloma participants.These participants were enrolled before the updated definition of multiple myeloma, Myeloma-defining events include ≥60% bone marrow plasmacytosis, serum-free light chain ratio≥100, &/or>1 focal lesion on magnetic resonance imaging. Between the time of initial enrollment in 2013, the definition of smoldering myeloma was changed to exclude participants with the listed myeloma defining events. The 10 participants in our cohort of high risk smoldering myeloma would be classified as having "full multiple myeloma" by today's definition.
  events | 10
High-risk Smoldering Multiple Myeloma by Programa de Estudio y Tratamiento de las Hemopatías Maligna [Count of Participants; unit: Participants] — High-risk is defined by immunoparesis ≥95% aberrant plasma cells on bone marrow aspirate flow cytometry Programa de Estudio y Tratamiento de las Hemopatías Malignas (PETHEMA). This is just one high risk criteria. Neither good nor bad for the participant.
  Participants | 36
Number of Participants with High-Risk Smoldering Multiple Myeloma (SMM) by Mayo Clinic 2008 [Count of Participants; unit: Participants] — High-risk is defined by a serum-free light chain ratio of 8 or 0.125 (Mayo Clinic 2008) or 2-3 of the following: serumMprotein >2 g/dL, involved to uninvolved free light chain ratio >20, or bone marrow plasmacytosis >20%. This is just one high risk criteria. Neither good nor bad for the participant.
  Participants | 8
Number of Participants with High-Risk Smoldering Multiple Myeloma (SMM) by Mayo Clinic 2018 [Count of Participants; unit: Participants] — These participants were enrolled before the updated definition of multiple myeloma, Myeloma-defining events include ≥60% bone marrow plasmacytosis, serum-free light chain ratio ≥100, and/or >1 focal lesion on magnetic resonance imaging. This is just one high risk criteria. Neither good nor bad for the participant.
  Participants | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Minimal Residual Disease (MRD)Negative Complete Response (CR) Per International Myeloma Working Group (IMWG) Criteria
Description: MRDnegative Complete Response (CR) per the IMWHG criteria is defined as absence of phenotypically aberrant clonal plasma cells by flow cytometry on bone marrow aspirates using the eight-color two tube approach with a minimum sensitivity of 1 in 10^5 nucleated cells or higher.
Time Frame: 8 months
Population: 54/55 participants are evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 54
percentage of participants | 70.4 [56.4 to 82.0]

2. Secondary Outcome: Percentage of Participants That Have Minimal Residual Disease (MRD)-Negative Complete Response (CR) for a Minimum of 1 Year
Description: Percentage of participants that have Minimal Residual Disease (MRD)-negative Complete Response (CR) for a minimum of 1 year estimated along with a 95% two-sided confidence interval. MRDnegative Complete Response (CR) is defined as absence of phenotypically aberrant clonal plasma cells by flow cytometry on bone marrow aspirates using the eight-color two tube approach with a minimum sensitivity of 1 in 10^5 nucleated cells or higher.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 54
percentage of participants | 63 [49.0 to 76.0]

3. Secondary Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 117 months and 1 day.
Population: 54/55 participants are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 54
Participants | 54

4. Secondary Outcome: Clinical Progression Free Survival
Description: Clinical progression was assessed by the International Myeloma Working Group Criteria for Multiple Myeloma. Progression is any one of the following: Increase of ≥25% from lowest response value in the following on 2 consecutive measurements: Serum M-component and/or (the absolute increase must be ≥0.5g/dl). The serum M-component increases of ≥1 gm/dl are sufficient to define relapse if starting M-component is ≥0.5g/dl. Urine M-component and/or (the absolute must be ≥200mg/24h. Only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain (FLC) levels. The absolute increase must be >10mg/dl. Bone marrow plasma cell percentage: the absolute % must be ≥10%. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in size of existing bone lesions or soft tissue plasmacytomas. Development of hypercalcemia that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: time from enrollment in the study until development of overt clinical multiple myeloma (end organ damage or myeloma-defining event) or death, up to 5 years
Population: 54/55 participants are evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 54
percentage of participants | 90.7 [71.0 to 97.2]

5. Secondary Outcome: Biochemical Progression Free Survival
Description: Biochemical progression free survival is defined as the time from enrollment in the study until development of overt clinical multiple myeloma (end organ damage or myeloma-defining event) or death, and progressive disease by International Myeloma Working Group (IMWG) criteria. Progression is any one of the following: Increase of ≥25% from lowest response value in the following on 2 consecutive measurements: Serum M-component and/or (the absolute increase must be ≥0.5g/dl). The serum M-component increases of ≥1 gm/dl are sufficient to define relapse if starting M-component is ≥0.5g/dl. Urine M-component and/or (the absolute must be ≥200mg/24h. Only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain (FLC) levels. The absolute increase must be >10mg/dl. Bone marrow plasma cell percentage: the absolute % must be ≥10%.
Time Frame: time from enrollment in the study until development of overt clinical multiple myeloma (end organ damage or myeloma-defining event) or death, and progressive disease by IMWG criteria, up to 5 years
Population: 54/55 participants are evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 54
percentage of participants | 76.6 [59.2 to 87.3]

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from partial response to disease progression. Response was assessed by the International Myeloma Working Group Criteria for Multiple Myeloma. Partial Response is ≥50% reduction if serum M-protein and reduction in 24-hour(h) urinary M-protein by ≥90% or to <200mg per 24h. If the serum and urine M-protein are unmeasurable, a ≥50% decrease in the difference between involved and uninvolved free light chain (FLC) levels is required in place of the M-protein criteria. Progression is any one of the following: Increase of ≥25% from lowest response value in the following on 2 consecutive measurements: Serum M-component and/or (the absolute increase must be ≥0.5g/dl). The serum M-component increases of ≥1 gm/dl are sufficient to define relapse if starting M-component is ≥0.5g/dl. Urine M-component and/or (the absolute must be ≥200mg/24h.
Time Frame: time from partial response to disease progression, up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-01

7. Secondary Outcome: Overall Response Rate
Description: Overall response is defined as the percentage of participants who have a partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR) defined by the International Myeloma Working Group Criteria for Multiple Myeloma out of all evaluable participants. PR is ≥50% reduction if serum M-protein and reduction in 24-hour(h) urinary M-protein by ≥90% or to <200mg per 24h. If the serum and urine M-protein are unmeasurable, a ≥50% decrease in the difference between involved and uninvolved free light chain (FLC) levels is required in place of the M-protein criteria. VGPR is serum and urine M-protein detectable by immunofixation but not on electrophoresis. CR is negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and ≥5% plasma cells in bone marrow. sCR is complete response plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
Time Frame: time measurement criteria are met for best response until the first date that recurrent or progressive disease is met, up to 5 years
Population: 54/55 participants are evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 54
percentage of participants
  Overall Response Rate | 100
  Partial Response | 5.5
  Very Good Partial Response | 18.5
  Complete Response | 0
  Stringent Complete Response | 75.9

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 117 months and 1 day.
Description: 54/55 participants are evaluable for adverse events.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 12/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=54)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Ear and labyrinth disorders - Other, Labyrinthitis (Ear and labyrinth disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal disorders - Other, Lower gastrointestinal (GI) Bleed (Gastrointestinal disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (2)
Lung infection (Infections and infestations) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=54)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Activated partial thromboplastin time prolonged (Investigations) | 3 (7)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 14 (46)
Alkaline phosphatase increased (Investigations) | 15 (27)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 16 (59)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 10 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Bloating (Gastrointestinal disorders) | 11 (11)
Blood bilirubin increased (Investigations) | 7 (26)
Blurred vision (Eye disorders) | 7 (7)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
CPK increased (Investigations) | 6 (8)
Cataract (Eye disorders) | 2 (3)
Chills (General disorders) | 4 (4)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 21 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Creatinine increased (Investigations) | 10 (29)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 29 (55)
Dizziness (Nervous system disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 15 (15)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Edema limbs (General disorders) | 15 (23)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye disorders - Other, Stye-right upper lid (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 32 (45)
Fever (General disorders) | 10 (12)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Flu like symptoms (General disorders) | 5 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 17 (18)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Haptoglobin decreased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 11 (16)
Heart failure (Cardiac disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (13)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (14)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 7 (7)
Hypernatremia (Metabolism and nutrition disorders) | 10 (22)
Hypertension (Vascular disorders) | 9 (10)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (43)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (14)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (16)
Hyponatremia (Metabolism and nutrition disorders) | 3 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (19)
Infections and infestations - Other, Blood (Infections and infestations) | 1 (2)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 4 (4)
Infections and infestations - Other, Herpes Simplex Virus (Shingles) (Infections and infestations) | 1 (1)
Infections and infestations - Other, Tick bite (Infections and infestations) | 1 (1)
Infections and infestations - Other, nausea and vomiting for one time with diarrhea (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Injection site reaction (General disorders) | 13 (22)
Insomnia (Psychiatric disorders) | 19 (22)
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (3)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Libido decreased (Reproductive system and breast disorders) | 1 (1)
Localized edema (General disorders) | 3 (3)
Lung infection (Infections and infestations) | 10 (10)
Lymphocyte count decreased (Investigations) | 18 (144)
Lymphocyte count increased (Investigations) | 1 (1)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Fasciculation (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, muscle cramp, right calf -intermittent (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (21)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 18 (22)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, BCC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Liver and pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous system disorders - Other, Myokimia (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 18 (77)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 1 (1)
Pain (General disorders) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 4 (5)
Paresthesia (Nervous system disorders) | 4 (4)
Paronychia (Infections and infestations) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (19)
Phlebitis (Vascular disorders) | 11 (14)
Platelet count decreased (Investigations) | 19 (73)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (12)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 35 (55)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Infiltrate (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5)
Skin and subcutaneous tissue disorders - Other, Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Right knee Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Skin nodules (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Nodules (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Spasticity (Nervous system disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 11 (11)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 14 (18)
Urinary frequency (Renal and urinary disorders) | 4 (5)
Urinary tract infection (Infections and infestations) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 18 (97)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT01572480/Prot_SAP_002.pdf
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT01572480/ICF_003.pdf